CLINICAL TRIAL: NCT07096739
Title: Tolerance and Acceptance of a High Protein Nutrition Shake in Individuals Treated With the GLP-1 Receptor Agonist Semaglutide: a Single Arm, Open Label Study
Brief Title: Tolerance of a High Protein Nutrition Shake in Individuals on GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kate Farms Inc (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INQUIS2025
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: GLP-1 Concentration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Subjects will consume the study product daily for 1 week.
  Interventions: Dietary Supplement: High protein shake

INTERVENTIONS:
Dietary Supplement: High protein shake — Subjects in this study will consume the study product for 1 week. Participants will record GI symptoms over the past 24h on 3 days during the week prior to the intervention, and on days 3, 5, and 7 during the intervention. On the first day, overnight fasted participants will be given the product and symptoms will be followed for 2h. 24h dietary recalls will be collected at the beginning and end of the 7-day treatment period.

SUMMARY:
Determine if consuming a high protein nutrition shake reduces gastrointestinal symptoms associated with semaglutide injections.

DETAILED DESCRIPTION:
This study investigates the tolerability of a shake specifically designed to reduce GI side effects in individuals being treated with the GLP-1 agonist semaglutide. The study uses a single-arm, open label design where subjects will consume the study product daily for 1 week. Participants will record GI symptoms over the past 24h on 3 days during the week prior to the intervention, and on days 3, 5 and 7 during the intervention

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals aged 18-75 years, inclusive
* BMI >27.0kg/m²
* Taking semaglutide injections (Ozempic or Wegovy) as prescribed (eg. weekly), for at least 4 weeks prior to screening
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP
* Subjects must have an active e-mail address, daily access to an electronic device (e.g. computer, laptop, tablet, smart phone) and internet, and understand how to complete the daily electronic diary daily

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria
2. Use of a compounded GLP-1 agonist
3. Reported history of metabolic (including type 1 and type 2 diabetes mellitus), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, psychiatric disorders, or any other medical conditions that, in the judgment of the Principal Investigator, increase the risk to the subject or others or may affect results
4. Hospital admission for major trauma, or major medical or surgical event, as judged by the Principal Investigator, within 6 months of screening
5. Use of medications such as, but not limited to, hypoglycemic agents, systemic steroids, antipsychotics, or any others that increase the risk to the subject or others or may affect results, as judged by the Principal Investigator
6. Known intolerance, sensitivity, or allergy to any ingredients in the study test products
7. Self-reported pregnancy or breastfeeding or less than 6 weeks postpartum
8. Long term treatment with another investigational drug or other intervention within the last 30 days
9. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Composite GI symptoms score (CSS) | 7 days
  Comparison of the composite GI symptom scores (CSS) recorded during the 7day intervention period with those recorded during the 3-day baseline period.

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis Clinical Research, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No